CLINICAL TRIAL: NCT03444077
Title: Impact of a Prehospital Discrimination Between Trauma Patients With or Without Early Acute Coagulopathy of Trauma and the Need for Damage Control Resuscitation : a Multicenter Randomized Phase II Trial.
Brief Title: Impact of a Prehospital Identification of Trauma Patients in Need for Damage Control Resuscitation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Martin L Tonglet, MD, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: STTTOPPP the bleeding trial
Record Dates: First submitted 2018-02-18; First posted 2018-02-23 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Trauma; Coagulopathy; Hemorrhage; Emergencies
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders; Hemorrhage; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The patients allocated in the control group will be managed as recommended in the local guidelines and protocols. As the trial involves participating centers with different prehospital and hospital realities and local practices, the control group will reflect a wide panel of levels of care and will not be limited to a unique approach.
  Interventions: Diagnostic Test: Regular care; Other: Regular Care
- Intervention group (Experimental): Patients will be classified in two categories regarding their TICCS value. Patients with TICCS ≥ 10 will be classified as in need for DCR; while patients with TICCS < 10 will be classified as not in need for DCR.
  TICCS < 10 This subgroup will be considered without a need for DCR and without coagulopathy. There will not be any activation of the DCR components (no phone contact to the blood bank, to the surgical team, no prehospital transfusion). There will be any prehospital treatment/prevention of the hyperfibrinolysis using Tranexamic acid (TXA). Crystalloids infusion will be allowed.
  TICCS ≥ 10 This subgroup will be considered with a need for DCR and with coagulopathy. They will be treated using the STTTOPPP the bleeding protocol.
  Interventions: Diagnostic Test: Use of the Trauma Induced Coagulopathy Clinical Score (TICCS) as a diagnostic tool.; Other: STTTOPPP the bleeding

INTERVENTIONS:
Diagnostic Test: Use of the Trauma Induced Coagulopathy Clinical Score (TICCS) as a diagnostic tool. — The TICCS will be calculated on the site of injury for the patients taken in charge in the intervention group. Those patients will be classified in two categories regarding their TICCS value. Patients with TICCS ≥ 10 will be classified as in need for DCR; while patients with TICCS < 10 will be classified as not in need for DCR.
  Arms: Intervention group
Diagnostic Test: Regular care — Patients from the control group will be evaluated by clinicians using the local usual clinical Tools.
  Arms: Control group
Other: STTTOPPP the bleeding — * Surgical team pre-activation
  * Trauma team pre-activation
  * Transfusion team pre-activation
  * Tranexamic acid (administration of 1 gram of TXA if documented hyperfibrinolysis)
  * O negative RBC transfusion as soon as possible
  * Plasma and Platelets transfusion as soon as possible
  * Permissive hypotension (restrictive use of crystalloids: no more than 500 milliliters before definitive control of the bleeding is achieved)
  * Prophylaxis (initiate antithrombotic prophylaxis as soon as the bleeding is under control and coagulation tests are normal, first evaluation before the 24th hour after trauma)
  Arms: Intervention group
Other: Regular Care — Regular local pre-hospital care.
  Arms: Control group

SUMMARY:
Early identification of trauma patients in need for Damage Control Resuscitation (DCR) has potential to be beneficial for general emergency units that are not expected to be ready for this rare situation 24 hours per day, 7 days per week. It could also be useful for high performing trauma centers to identify such patients earlier and be able to provide earlier adequate treatment.

By contrast, initiation of DCR in patients who do not require this aggressive therapy may negatively affect their survival. An early identification of patients who do not require DCR would probably be beneficial (impact on cost-effectiveness and on patients' survival).

The evidence of the Trauma Induced Coagulopathy Clinical Score (TICCS) accuracy has been evaluated in several studies but the potential effect of its use on patient outcomes needs to be evaluated. There has never been any evaluation of the impact of a prehospital discrimination of trauma patients with or without the need for DCR.

The primary objective of this study is to evaluate the impact on mortality of a prehospital discrimination between trauma patients with or without a potential need for DCR. Secondary objectives include evaluation of the feasibility of such discrimination and its impact on cost-effectiveness. We hypothesize that the information will lead to improved quality of care with reduced mortality and morbidity.

DETAILED DESCRIPTION:
The trial will be designed as randomized phase II clinical trial with comparison of the experimental protocol (prehospital discrimination using the TICCS) against the standard of care. Patients will be allocated in a 1:1 ratio in two groups: the intervention group will benefit from a prehospital evaluation using the TICCS and from a specific treatment protocol regarding the TICCS value. The control group will benefit from the standard local care.

The trial will involve several participating prehospital and hospital teams across Belgium.

Control and intervention group will only differ in the management of potential bleeding and coagulopathy. All patients will benefit from the recommended level of care regarding their situation, including airway management, Traumatic Brain Injury (TBI) management, control of external bleeding, cervical spine and extremities immobilization if needed …

Control group The patients allocated in the control group will be managed as recommended in the local guidelines and protocols. As the trial involves participating centers with different prehospital and hospital realities and local practices, the control group will reflect a wide panel of levels of care and will not be limited to a unique approach.

Intervention group The TICCS will be calculated on the site of injury for the patients taken in charge in the intervention group. Those patients will be classified in two categories regarding their TICCS value. Patients with TICCS ≥ 10 will be classified as in need for DCR; while patients with TICCS < 10 will be classified as not in need for DCR.

TICCS < 10 This subgroup will be considered without a need for DCR and without coagulopathy. There will not be any activation of the DCR components (no phone contact to the blood bank, to the surgical team, no prehospital transfusion). There will be any prehospital treatment/prevention of the hyperfibrinolysis using Tranexamic acid (TXA). Crystalloids infusion will be allowed. All patients will benefit from the recommended level of care regarding their situation (airway, TBI …), including trauma team activation if locally recommended.

TICCS ≥ 10

This subgroup will be considered with a need for DCR and with coagulopathy. They will be treated using the STTTOPPP the bleeding protocol. The STTTOPPP the bleeding protocol is the acronym for:

* Surgical team pre-activation
* Trauma team pre-activation
* Transfusion team pre-activation
* Tranexamic acid (administration of 1 gram of TXA if documented hyperfibrinolysis)
* O negative Red Blood Cells (RBC) transfusion as soon as possible
* Plasma and Platelets transfusion as soon as possible
* Permissive hypotension (restrictive use of crystalloids: no more than 500 milliliters before definitive control of the bleeding is achieved)
* Prophylaxis (initiate antithrombotic prophylaxis as soon as the bleeding is under control and coagulation tests are normal, first evaluation before the 24th hour after trauma)

Data will be collected locally in each participating center and will be anonymously recorded on the trial website by the local Principal Investigator or his research assistant. The website has been designed to avoid incomplete data, will give feedbacks (about the number of patients included) to this respective centers every six months. The participating centers will only have access to their own center database. The trial coordination team will have access to the whole database and will not be able to record or change any data. After one year of inclusion and in the end of the 24 months period of inclusion, data will be extracted for interim and final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Prehospital intervention of paramedical or medical team involved in the present trial
* Admission in a hospital involved in this trial

Exclusion Criteria:

* Spontaneous admission without prehospital intervention
* Penetrating trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Seven days mortality | seven days
  Overall mortality

SECONDARY OUTCOMES:
Thirty days mortality | Thirty days
  Overall mortality
Hospital length-of-stay | Thirty days
  Overall hospital length-of-stay
Blood products transfusion | Thirty days
  Total number of blood products transfused during the hospitalization (units)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Ghuysen, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (4):
- Belgium (4):
  - Centre Hospitalier Universitaire St Pierre, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Réseau hospitalier de Jolimont, La Louvière
  - Centre Hospitalier Universitaire de Liège, Liège

IPD SHARING:
Plan to Share IPD: No